CLINICAL TRIAL: NCT00591643
Title: Adrenal Scans With Radioiodine-Labeled Norcholesterol (NP-59)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 77-030
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Adrenal Tumors; Adrenal Malignancies; Abnormal Hormonal Secretions; Electrolytes Abnormalities
Keywords: Adrenal tumors; Adrenal malignancies; abnormal hormonal secretions; electrolytes abnormalities; Imaging; Scanning; tumor localization
MeSH Terms: conditions — Adrenal Gland Neoplasms | interventions — X-Rays; Adosterol

ARMS (1):
- Imaging, Adrenal acans & Radiation (Experimental)
  Interventions: Procedure: Imaging, Adrenal acans; Radiation: (NP-59)

INTERVENTIONS:
Procedure: Imaging, Adrenal acans — The patient will be given 5 drops of saturated solution of potassium iodide daily for 2 days prior to the study and will continue for 5 to 7 days later to minimize the radiation dose to the thyroid gland. One to 2 mCi of I 131 1,6-beta-iodomethyl-19-norcholesterol (NP-59) in 10% ethanol, 0.23% polysorbate 80 and 0.9% NaCl will be given intravenously slowly over 1-5 minutes. Anterior and posterior images of the adrenal area will be obtained 72 and 96 hours later. Additional images will be made if indicated. Each image would require 30 minutes carried out in the nuclear medicine laboratory. To verify the exact location of the adrenal glands, renal scan with 99m Tc DTPA or Mag 3 (routine nuclear medicine radiopharmaceuticals) will also be obtained whenever indicated. In some patients, dexamethasone suppression will be carried out to improve the specificity of NP 59 diagnosis for autonomous hormonal secretions by the adrenal tumors.
Radiation: (NP-59) — One to 2 mCi of I 131 1,6-beta-iodomethyl-19-norcholesterol (NP-59) in 10% ethanol, 0.23% polysorbate 80 and 0.9% NaCl will be given intravenously slowly over 1-5 minutes.

SUMMARY:
The purpose of this study is to find out if your adrenal glands are normal or abnormal. This can be determined by whether or not your adrenal gland concentrates more of a labeled building block of adrenal hormone, norcholesterol. This labeled material had been used as an investigative diagnostic tool for imaging adrenal glands for many years with success in our hands. This is a diagnostic procedure. CT, MRI and Ultrasound can determine the size and presence or absence of tumor but cannot assess the function of the adrenal glands. To determine hormone concentrations from blood samples would involve more invasive catherization.

DETAILED DESCRIPTION:
To investigate the feasibility of using NP-59 to localize adrenal tumors and assess their functions under the influence of pharmacological manipulations.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical and laboratory suspicions of hypersecretion of adrenal cortical hormones

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 1977-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To investigate the feasibility of using NP-59 to localize adrenal tumors and assess their functions under the influence of pharmacological manipulations. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Pandit-Taskar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering web site — http://www.mskcc.org